CLINICAL TRIAL: NCT04111744
Title: Preoperative Excercise Training for Patients Undergoing Coronary Artery Bypass Graft Surgery- A Prospective Randomized Trial
Brief Title: Preoperative Excercise Training for Patients Undergoing Coronary Artery Bypass Graft Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kerckhoff Klinik (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: PRECAB
Record Dates: First submitted 2018-03-21; First posted 2019-10-01 (Actual); Last update posted 2019-10-01 (Actual); Status verified 2019-09

CONDITIONS: Coronary Artery Disease; Physical Activity; Coronary Artery Bypass Graft Surgery
Keywords: Coronary Artery Bypass Graft Surgery; Physical Activity; Coronary Artery Disease; Physical Training
MeSH Terms: conditions — Coronary Artery Disease; Motor Activity

STUDY DESIGN:
Intervention Model Description: Patients enrolled to the study were randomised in a Treatment and a control Group
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Training Group (Experimental): Preoperative Exercise Training Optimal medical therapy,
  Interventions: Other: Preoperative Exercise Training; Other: Optimal medical therapy
- Control Group (Other): Optimal medical therapy, inactive control group
  Interventions: Other: Optimal medical therapy

INTERVENTIONS:
Other: Preoperative Exercise Training — Patients undergoing CABG and randomized to the Training Group complete six sessions of aerobic endurance training prior CABG surgery
  Arms: Training Group
Other: Optimal medical therapy — Standard medication for stable CAD

SUMMARY:
Patients (pts) with stable coronary artery disease (CAD) requiring coronary artery bypass graft surgery (CABG) may be physically inactive during the waiting period to avoid further risks. Aim of this study is to investigate the feasibility and safety of a preoperative aerobic exercise training in these pts during the waiting period and to analyze its effects on pre-, peri and postoperative outcomes

DETAILED DESCRIPTION:
Pts with stable coronary artery disease (CAD) and indication for elective CABG will be prospectively randomized into a preoperative training group (TG) or a non active control group (CG). Pts in TG have to perform six sessions of aerobic endurance training within two weeks prior to CABG. The following investigations will be performed at baseline, one day before surgery and at the beginning and at the end of cardiac rehabilitation: a maximal symptom limited ergospirometry, assessment of endothelial function (analysing the reactive hyperaemic index (RHI) via a finger-tonometry), assessment of quality of life (QoL) using the MacNew Heart Disease Questionnaire, laboratory testing of ischemic and inflammatory Parameters. Baseline, peri- and postoperative characteristics will be collected.

ELIGIBILITY:
Inclusion Criteria:

* stable Angina
* indication for elective CABG surgery
* functional capacity > 50 watts
* willingness to participate in the study

Exclusion Criteria:

* unstable Angina
* comorbidities precluding performance of aerobic exercise training (e.g. neurological disorders, orthopedic disorders etc)
* functional Status NYHA IV
* relevant ventricular arrhythmias
* hemodynamic significant heart valve disease
* myocarditis
* cardiomyopathies
* left main coronary artery disease > 50%
* peripheral obstructive disease (Fontaine > IIb)
* reduced life expectancy < 12 months
* CABG surgery during the last six months
* participation in another trial

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 203 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Cardiopulmonary fitness | Baseline, prior surgery on hospital admission day, hospital discharge day ( postoperative day 7-14) , after 3 weeks of cardiac rehabilitation
  Change of maximal Oxygen consumption
Endothelial function | Baseline, prior surgery on hospital admission day, hospital discharge day (postoperative day 7-14), after 3 weeks of cardiac rehabilitation
  Change of Reactive hyperemic index (RHI)

SECONDARY OUTCOMES:
Length of hospital stay (LoS) | Within the acute care period
  Duration of hospital stay in days
Length of ventilation | Within the acute care period
  Duration of Ventilation in minutes
Functional capacity | Baseline, prior surgery on hospital admission day, hospital discharge day(postoperative day 7-14), , after 3 weeks of cardiac rehabilitation
  Change of 6-minute walk test
Arterial stiffness | Baseline, prior surgery on hospital admission day, hospital discharge day(postoperative day 7-14), , after 3 weeks of cardiac rehabilitation
  Changes in arterial pulse wave analysis
Quality of life Questionnaire 1 | Baseline, prior surgery on hospital admission day, hospital discharge day(postoperative day 7-14), , after 3 weeks of cardiac rehabilitation
  Changes in MacNew (Heart Disease Health-related Quality of Life-) Questionnaire questionaire
Quality of life Questionnaire 2 | Baseline, prior surgery on hospital admission day, hospital discharge day(postoperative day 7-14), , after 3 weeks of cardiac rehabilitation
  Changes in Hospital Anxiety and Depression Scale (HADS) questionnaire: The HADS is a fourteen item scale that generates ordinal data.Each item on the questionnaire is scored from 0-3 and this means that a person can score between 0 and 21 for either anxiety or depression.
Quality of life Questionnaire 3 | Baseline, prior surgery on hospital admission day, hospital discharge day(postoperative day 7-14), , after 3 weeks of cardiac rehabilitation
  Changes in Mobility and Self-supply (MOSES) questionnaire
Ischemic blood marker 1 | Baseline, prior surgery on hospital admission day, hospital discharge day(postoperative day 7-14), , after 3 weeks of cardiac rehabilitation
  High Sensitive Troponin (hs-Trop)
Ischemic blood marker 2 | Baseline, prior surgery on hospital admission day, hospital discharge day(postoperative day 7-14), , after 3 weeks of cardiac rehabilitation
  Creatine kinase (CK) U/L
Ischemic blood marker 3 | Baseline, prior surgery on hospital admission day, hospital discharge day(postoperative day 7-14), , after 3 weeks of cardiac rehabilitation
  Creatine Kinase-MB (CK-MB) U/L
Ischemic blood marker 4 | Baseline, prior surgery on hospital admission day, hospital discharge day(postoperative day 7-14), , after 3 weeks of cardiac rehabilitation
  Lactate dehydrogenase (LDH) U/L
Ischemic blood marker 5 | Baseline, prior surgery on hospital admission day, hospital discharge day(postoperative day 7-14), , after 3 weeks of cardiac rehabilitation
  glutamic oxaloacetic transaminase (GOT) U/L
Ischemic blood marker 6 | Baseline, prior surgery on hospital admission day, hospital discharge day(postoperative day 7-14), , after 3 weeks of cardiac rehabilitation
  glutamate pyruvate transaminase (GPT) U/L
Ischemic blood marker 7 | Baseline, prior surgery on hospital admission day, hospital discharge day(postoperative day 7-14), , after 3 weeks of cardiac rehabilitation
  copeptin U/L
Inflammatory blood marker 1 | Baseline, prior surgery on hospital admission day, hospital discharge day(postoperative day 7-14), , after 3 weeks of cardiac rehabilitation
  C-reactive protein (CRP) U/L
Inflammatory blood marker 2 | Baseline, prior surgery on hospital admission day, hospital discharge day(postoperative day 7-14), , after 3 weeks of cardiac rehabilitation
  Leucozytes 10³/µL
Inflammatory blood marker 3 | Baseline, prior surgery on hospital admission day, hospital discharge day(postoperative day 7-14), , after 3 weeks of cardiac rehabilitation
  Interleukine-6 (IL-6) pg/mL
Number of patients with a Clinical Event | Baseline, prior surgery on hospital admission day, hospital discharge day(postoperative day 7-14), , after 3 weeks of cardiac rehabilitation
  Atrial fibrillation documented by electrocardiogram (ECG)
Number of patients with a Pulmonary clinical event | Baseline, prior surgery on hospital admission day, hospital discharge day(postoperative day 7-14), , after 3 weeks of cardiac rehabilitation
  Pleural effusion, pulmonary infection or other pulmonary disorder with Need for treatment
Number of patients with a Cardiovascular event | after 30 days and 12 months
  Revascularization, re-CABG, rehospitalization due to unstable angina, myocardial infarction
Number of patients with a Cerebrovascular event | after 30 days and 12 months
  TIA, stroke

CONTACTS AND LOCATIONS:
Overall Officials: Claudia Walther, MD, Principal Investigator — Kerckhoff Clinic; Heike Baumgarten, MD, Principal Investigator — Kerckhoff Clinik
Locations (1):
- Kerckhoff Klinik, Bad Nauheim, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Steinmetz C, Bjarnason-Wehrens B, Baumgarten H, Walther T, Mengden T, Walther C. Prehabilitation in patients awaiting elective coronary artery bypass graft surgery - effects on functional capacity and quality of life: a randomized controlled trial. Clin Rehabil. 2020 Oct;34(10):1256-1267. doi: 10.1177/0269215520933950. Epub 2020 Jun 16. PMID 32546065